CLINICAL TRIAL: NCT01094457
Title: Effects of Intensive Antiplatelet Therapy for Patients With Clopidogrel Resistance After Coronary Stent Implantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Yaling Han, vice president, Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 825004-5
Record Dates: First submitted 2010-03-26; First posted 2010-03-29 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Acute Coronary Syndromes; Percutaneous Coronary Intervention; Clopidogrel Low Responsiveness
Keywords: antiplatelet therapy; clopidogrel low responsiveness; acute coronary syndromes; percutaneous coronary intervention; cilostazol
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Aspirin; Clopidogrel; Cilostazol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard group (Active Comparator): patients in this group received standard dual antiplatelet therapy, i.e. aspirin 300mg/d and clopidogrel 75mg/d
  Interventions: Drug: aspirin, clopidogrel
- intensive group (Experimental): patients in this group received intensive antiplatelet therapy and the regimen can be adjusted according to results of platelet aggregation function test by LTA
  Interventions: Drug: aspirin, clopidogrel, cilostazol

INTERVENTIONS:
Drug: aspirin, clopidogrel — patients in the standard group received standard dual antiplatelet therapy: aspirin 300mg/d for 30 days followed by 100mg/d indefinitely, clopidogrel 75mg/d for at least 1 year
  Arms: standard group
Drug: aspirin, clopidogrel, cilostazol — Firstly,all patients in this group were received aspirin 300mg/d and clopidogrel 150mg/d for 3 days. Then a platelet aggregation function test was performed. The regimen will lasted for another 27 days if patients were judged as responsive to current clopidogrel dose. Patients still with clopidogrel resistance were then randomly assigned to receive clopidogrel 75mg/d plus cilostazol 100mg, twice per day or clopidogrel 150mg/d plus cilostazol 50mg, twice per day for 27 days. At 30-day, a repeat platelet aggregation function test wil performed for all patients. Then a standard dual antiplatelet regimen with aspirin 100mg/d indefinitely and clopidogrel 75mg/d for at least 1 year will be prescribed for all patients.
  Arms: intensive group

SUMMARY:
Clopidogrel resistance (CR) or low-responsiveness is associated with increased risk of ischemic events and can be detected by laboratory tests. This multicenter, randomized study is aimed to explore the efficacy and safety of intensive antiplatelet therapy (i.e. double clopidogrel maintenance dose and/or additional cilostazol)for patients with CR after coronary stenting.

ELIGIBILITY:
Inclusion Criterial:

* aged 35 to 75 years
* acute coronary syndromes
* underwent successful coronary stent implantation
* informed consent

Exclusion Criteria:

* contraindications to antiplatelet therapy
* history of intracranial bleeding
* known bleeding disorders
* severe liver or kidney disease
* pregnancy
* left main coronary artery disease
* planned non cardiac surgery within 1 year
* end stage of other serious disease with life expectancy less than 1 year
* heart failure with NYHA grade 3 to 4

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2009-03; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Major ischemic cardiovascular events | 1 year
  defined as a composite of cardiac death, myocardial infarction or stroke

SECONDARY OUTCOMES:
Stent thrombosis | 1 year
  according to ARC definition
major adverse cardiac and cerebral events(MACCE) | 1 year
  defined as a composite of cardiac death, myocardial infarction, target vessel revascularization or stroke
Hemorrhagic events | within 1 year
  according to TIMI bleeding definition
reduction in ADP induced platelet aggregation | 30 days
  assessed by LTA (Packs-4 Aggregometer, Helena labs, Beaumont, Texas)

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, MD, Principal Investigator — Shenyang Northern Hospital
Locations (3):
- China (3):
  - 463 Hospital of PLA, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Shenyang Northern Hospital, Shenyang, Liaoning